CLINICAL TRIAL: NCT04367753
Title: Predictive Factors for the Results of Epiphysiodesis in Limb Length Discrepancy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 202PI078
Record Dates: First submitted 2020-04-27; First posted 2020-04-29 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Limb Length Discrepancy
Keywords: Epiphysiodesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fulfilled contract: The contract before the epiphysiodesis has been fulfilled with the wanted limb length at the final analysis
- Failed contract: The contract before the epiphysiodesis hasn't been fulfilled with the wanted limb length at the final analysis

SUMMARY:
Several techniques exist for epiphysiodesis in limb length discrepancy with different results. Most of the time the results are disappointing for this functional surgery.

The aim of this study is understanding the reasons of the failures by analyzing the different steps of the medical care.

The patients will be distributed in two groups : "fulfilled contract" and "failed contract" The differences between the two groups will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with limb length discrepancy who had epiphysiodesis surgery

Exclusion Criteria:

* Missing x-rays
* missing data
* bone growth not achieved

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All minors with limb length discrepancy who had epiphysiodesis surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Limb length discrepancy before surgery | 3 months
Bones length | 3 months
Predictive bone growth | 3 months
Time limit between consultation and surgery | 3 months
Screw position in physis | 3 months
Bone age at the time of surgery | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Mathias KIRSCH, Principal Investigator — CHU Hôpital d'Enfants Nancy
Locations (1):
- CHU Hopitâl d'Enfants, Nancy, Lorraine, France

IPD SHARING:
Plan to Share IPD: Undecided